CLINICAL TRIAL: NCT05589285
Title: Outcomes of Autologous Whole Blood Injection for the Treatment of Plantar: A Randomized Controlled Trial.
Brief Title: Outcomes of Autologous Whole Blood Injection for the Treatment of Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Wafa Al Baluki, Consultant foot and ankle orthopaedics surgeon, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MREC 2864
Record Dates: First submitted 2022-10-10; First posted 2022-10-21 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Plantar Fascitis
Keywords: plantar fasciitis; Whole blood injection
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Chronic plantar fasciitis patients who will receive autologous whole blood injection.
  Interventions: Biological: Injection of autologous whole blood to the plantar fascia
- Control group (Sham Comparator): Chronic plantar fasciitis patients who will receive normal saline injection.
  Interventions: Device: Injection of normal saline to the plantar fascia

INTERVENTIONS:
Biological: Injection of autologous whole blood to the plantar fascia — Patients assigned in this group will have 2 ml of blood withdrawn from a peripheral vein, then mixed with 1 mL Lidocaine 2% for a total of 3mL volume in one syringe. The patient will be asked to lie down in the clinic bed, and the injection will be administered to the plantar fascia by the principal investigator using a sterile technique.
  Arms: Treatment group
Device: Injection of normal saline to the plantar fascia — This will be the control group receiving sham injection. Patients will have 2 ml of blood withdrawn from a peripheral vein for blinding proposes. They will be asked to lie down on the clinic bed, 1 ml of normal saline will be administered under sterile technique by the principal investigator. The blood that was withdrawn initially will be discarded.
  Arms: Control group

SUMMARY:
The aim of this study is to investigate the effectiveness of whole blood injection as a safe and effective method of treatment of chronic plantar fasciitis.

The hypothesis is that Autologous whole blood (AWB) injection is more effective than sham injections in the treatment of plantar fasciitis.

Participants will receive an autologous whole blood injection over the plantar fascia, and will be followed up to study the response.

Researchers will compare the effects with a control group who will receive normal saline injection.

DETAILED DESCRIPTION:
Research objectives and hypothesis. The aim of this study is to investigate the effectiveness of whole blood injection as a safe and effective method of treatment of chronic plantar fasciitis.

The hypothesis is that AWB injection is more effective than sham injections in the treatment of plantar fasciitis.

Study design and research methods:

1. Study design:Randomized prospective single blinded study
2. Primary and secondary endpoints:

   Patients will be followed 6, 12, 24 weeks, and 12 months after the injection to assess the effects and improvement of symptoms.

   The outcomes will be measured using different scales that reflects resolution of symptoms such us: Visual Analog Scale (VAS), Foot Function Index (FFI) Foot and Ankle Ability Measure (FAAM). All questionnaires will be translated to Arabic for Arabic speakers. Moreover, the thickness of the plantar fascia will be measured by ultrasound before and after treatment. The operator of the ultrasound is a foot and ankle consultant trained on operating ultrasound.
3. Study treatments or interventions. Patients with the diagnosis of chronic plantar fasciitis will be recruited to the clinic and asked to participate. The primary investigator and co-investigators will be responsible to explain the nature of the study and take a written informed consent prior to inclusion in the study.

Treatment method for group 1:

Patients assigned in this group will have 2 ml of blood withdrawn from a peripheral vein, then mixed with 1 mL Lidocaine 2% for a total of 3mL volume in one syringe. The patient will be asked to lie down in the clinic bed, and the injection will be administered to the plantar fascia by the principal investigator using a sterile technique.

Treatment method for group 2:

This will be the control group (placebo group). Patients will have 2 ml of blood withdrawn from a peripheral vein for blinding proposes. They will be asked to lie down on the clinic bed, 1 ml of normal saline will be administered under sterile technique by the principal investigator. The blood that was withdrawn initially will be discarded.

Blinding:

Participants will not be aware on the type of injection they received, as both groups will have their blood withdrawn, and the injection will be prepared and given behind a curtain. Blinding of the investigators during treatment administration is not possible as the color of the syringe will give away the type of injection. The type of injection the patient received will not be mentioned in the electronic patient record. Thus, during all the subsequent follow up visits the investigator will not know which treatment group the patient is in to prevent bias.

Post injection:

All patients will be on the conservative management protocol of physiotherapy and orthotics and they will be instructed to perform stretching exercises on daily basis and to record it in dairy. There will be no restrictions in activity. Patients will be instructed not to use NSAIDs.

Randomization:

Patients will be randomized into two groups with a ratio of 1:1 using a computer based randomization system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic plantar fasciitis (persistence of symptoms despite 12 weeks of conservative management)
* Age: adults patients more than 18 years
* Not having responded to primary conservative managements such as rest, shoe insoles, conventional physical therapy, exercise therapy, and nonsteroidal anti-inflammatory drugs (NSAIDs).

Exclusion Criteria:

1. Neurological or vascular insufficiencies in the painful heel
2. Osteomyelitis, fracture of the calcaneus
3. Recent infection in the treatment area, history of rheumatic diseases
4. Immunosuppressive therapy or coagulation disturbance and/or therapy, long-term treatment with corticosteroids
5. Previous heel surgery
6. Patient with diabetes mellitus,
7. Pregnancy
8. Received corticosteroid injection
9. Four weeks since the last anaesthetic injection, iontophoresis, ultrasound and
10. electromyostimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 12 months
  Visual Analog Scale (VAS) to assess the pain score from 0 (minimum) to 10 (maximum)
Foot Function Index | 12 months
  a questionnaire based index to assess the foot function (from 0% minimum to 100% maximum)
Foot and Ankle Ability Measure (FAAM) | 12 months
  a questionnaire based index to assess foot and ankle ability in various daily life activities.
Change in Plantar fascia thickness | before the treatment and 12 months after the treatment.
  Measurement of the change in plantar fascia thickness using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Wafa Al Baluki, Principal Investigator — Sultan Qaboos University Hospital
Locations (1):
- Sultan Qaboos Univeristy Hospital, Muscat, Oman